CLINICAL TRIAL: NCT06629233
Title: Tn-Miner: Technology for the Discovery of Tumor-specific Glycopeptide Immunotherapy Targets.
Brief Title: Evaluation of a Novel Technique for the Discovery of New, Tumor-specific Targets for the Deployment of Innovative Immunotherapeutics Against Cancer.
Acronym: Tn-Miner
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONZ-2023-0589; F2022/IOF-StarTT/089 (Other Grant/Funding Number: Industrial Research Fund (IOF, UGent))
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Estrogen Receptor Positive Breast Cancer
MeSH Terms: interventions — Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care tumor resection (Other)
  Interventions: Procedure: Tumor resection

INTERVENTIONS:
Procedure: Tumor resection — As the standard of care, estrogen receptor-positive breast tumors are surgically resected. From these resected tumors, small samples of both cancer tissue and healthy surrounding tissue will be analyzed using our patented Tn-Miner workflow to discover novel tumor-specific epitopes.

SUMMARY:
The goal of this interventional, prospective research on human bodily material is to discover new, cancer-specific molecular structures (i.e. glycopeptides) within surgically removed, estrogen receptor positive breast cancer tumors.

The main goal it aims to achieve is:

To discover tumor-specific targets, that allow the use of very potent immunotherapeutic drugs as treatment for solid tumors, such as estrogen receptor positive breast cancer. These new targets are very specific for cancer cells, meaning that virtually no healthy cells should be attacked by the treatment, resulting in less side effects.

Participants will undergo standard of care treatment, comprising surgical removal of the breast tumor. Part of these tissues will be used for this clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Minimally 18 years old
* Diagnosed with estrogen-receptor positive breast cancer
* This must be a primary tumor

Exclusion Criteria:

* Male
* Younger than 18 years old
* Previous history of other tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Discovery of new, tumor-specific, glycopeptide epitopes. | The patients are only involved during their standard of care surgery (one day). The discovered epitopes will not be shared with enrolled patients.
  The discovery of new antigens, comprising both glycan and peptide (=glycopeptide), on the outside of the plasma membrane of the breast cancer cells. These antigens should be absent on healthy cells. These new, glycopeptide antigens can be used as target for immunotherapeutics against cancer.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Maria Middelares, Ghent, East-Flanders
  - University Hospital Ghent, Ghent, East-Flanders